CLINICAL TRIAL: NCT01260389
Title: Pharmaceutical Care for COPD Study
Brief Title: Pharmaceutical Care for Chronic Obstructive Pulmonary Disease (COPD) Study.
Acronym: PHARMACOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/2010/587
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): Usual pharmacist care in patients with Chronic Obstructive Pulmonary Disease (COPD).
- pharmaceutical care intervention (Experimental): A pharmaceutical care intervention, focused at improving inhalation technique and drug adherence in patients with Chronic Obstructive Pulmonary Disease (COPD).
  Interventions: Behavioral: pharmaceutical care intervention

INTERVENTIONS:
Behavioral: pharmaceutical care intervention — Pharmaceutical care intervention, focused at improving inhalation technique and drug adherence in patients with Chronic Obstructive Pulmonary Disease (COPD).
  Arms: pharmaceutical care intervention

SUMMARY:
This study would like to test the hypothesis that a pharmaceutical care intervention would result in an improved drug adherence and inhalation technique in Chronic Obstructive Pulmonary Disease (COPD) patients over a 3 month-period.

DETAILED DESCRIPTION:
Effective pharmacologic management of Chronic Obstructive Pulmonary Disease (COPD) not only involves prescription of recommended medicines by the physician, but also implies correct use of the prescribed medication by the patient (ie, good drug adherence and correct inhalation technique). Community pharmacists could help to improve the latter aspect, by delivering pharmaceutical care. The present randomised controlled trial will study the hypothesis that a pharmaceutical care intervention would result in an improved drug adherence and inhalation technique in COPD patients over a 3 month-period.

ELIGIBILITY:
Inclusion Criteria:

* daily use of Chronic Obstructive Pulmonary Disease (COPD)-medication: (Global initiative for chronic Obstructive Lung Disease: GOLD stadia I-IV)
* 50 years of age or older
* smoking history of at least 10 pack-years

Exclusion Criteria:

* having asthma
* analphabetism

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 734 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
inhalation technique baseline | baseline
  Inhalation technique with Chronic Obstructive Pulmonary Disease (COPD) controller medication at baseline.
inhalation technique 1 month | after 1 month
  Inhalation technique with Chronic Obstructive Pulmonary Disease (COPD) controller medication after 1 month.
inhalation technique 3 months | after 3 months
  Inhalation technique with Chronic Obstructive Pulmonary Disease (COPD) controller medication after 3 months.
drug adherence | after 3 months
  Adherence to Chronic Obstructive Pulmonary Disease (COPD) controller medication after 3 months.

SECONDARY OUTCOMES:
health status | baseline
  Health status, measured by:
  the Chronic Obstructive Pulmonary Disease (COPD) Assessment Test, Medical Research Council (MRC) Dyspnoea Scale and Euro Quality of Life (EQ-5D) questionnaire.
health status | after 1 month
  Health status, measured by:
  the COPD Assessment Test, MRC Dyspnoea Scale.
health status | after 3 months
  Health status, measured by:
  the COPD Assessment Test, MRC Dyspnoea Scale and EQ-5D questionnaire.
exacerbations | after 3 months
  Frequency of exacerbations measured over a 3 month period.
Emergency Room visits and hospitalizations. | after 3 months
  Frequency of Emergency Room (ER) visits and hospitalizations measured over a 3 month period.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Brusselle, M.D., Ph.D., Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Ghent University, Ghent
  - Centre Hospitalier Universitaire du Sart Tilman, Liège

REFERENCES:
- See also: Related Info — http://www.uzgent.be